CLINICAL TRIAL: NCT02667574
Title: Phase II Study Evaluating the Interest of Vismodegib as Neo-adjuvant Treatment of Basal Cell Carcinoma (BCC)
Brief Title: Study Evaluating the Interest of Vismodegib as Neo-adjuvant Treatment of Basal Cell Carcinoma (BCC)
Acronym: VISMONEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013_36; 2013-004338-13 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; surgery; stage; vismodegib
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label (Other): Enrolled patients will receive continuous once-daily oral dosing of Vismodegib at a dosage of 150 mg per administration (in accordance with the product SmPC). One cycle of therapy will be defined as 28 days of treatment. The treatment will be renewed once a month depending on the product tolerance
  Interventions: Drug: ERIVEDGE

INTERVENTIONS:
Drug: ERIVEDGE
  Other Names: VISMODEGIB

SUMMARY:
Open-label, non-comparative, multicenter, phase II study of Vismodegib in patients with locally advanced BCC.

DETAILED DESCRIPTION:
Enrolled patients will receive continuous once-daily oral dosing of Vismodegib at a dosage of 150 mg (in accordance with the product SmPC) per administration. One cycle of therapy will be defined as 28 days of treatment. The treatment will be renewed once a month depending on the product tolerance.

The trial will consist of a Screening Period (Day -28 to -1), a Treatment Period (Day 1 to BOR), one End of Treatment Visit, one Surgery Visit and 8 Safety Follow-Up Visits after the last dose of Vismodegib (+/- 5 days). Day 1 of the study will be defined as the first day a patient receives Vismodegib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with BCC, which surgery stage is A, B or C (cf. Appendix 3: Definition of surgery stages), with a diameter ≥ 3cm in zones at intermediate risk of tumor recurrence and a BCC with a diameter of ≥ 2 cm in the zones at higher risk of tumor recurrence. According to the HAS recommendations, two zones are taken into consideration:

   * Zones at intermediate risk of tumor recurrence: forehead, cheek, chin, neck and scalp
   * Zones at higher risk of tumor recurrence: nose and periorificial sites of the cephalic extremity
2. The decision to include the patient in this study should be taken during the Pluridisciplinary Committee Meeting (RCP). During this RCP, the radiotherapy should be considered as an inadequate treatment. (If the radiotherapist is absent during the meeting, his opinion should be documented in the patient's medical record).
3. Written informed consent
4. Age ≥ 18 years old
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0, 1, or 2
6. At least one histologically confirmed lesion...
7. Patients with Gorlin syndrome may enroll in this study but must meet the other inclusion criteria
8. Patients with measurable and/or non-measurable disease (as defined by RECIST, v1.1)
9. Adequate organ function, as evidenced by the following laboratory results:

   * Hemoglobin > 8.5 g/dL
   * Granulocyte count ≥ 1000/μL
   * Platelet count ≥ 75,000/μL
   * Aspartate transaminase (AST ) and alanine transaminase (ALT) ≤ 3 × upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 × ULN or within 3 × ULN for patients with documented Gilbert syndrome
10. Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
11. Women of childbearing potential must use one highly-effective method of contraception and one barrier method of contraception during treatment and for 24 months after the final dose. Highly-effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (e.g., implants, injectables, or intra-uterine devices; refer to Appendix 8 for more details). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, and postovulation methods] and withdrawal are not acceptable methods of contraception.).
12. For male patients with female partners of childbearing potential, agreement top use a condom with spermicide, even after vasectomy, during sexual intercourse with partners while being treated with Vismodegib and for two months after completion of study treatment
13. For male patients, agreement not to donate semen during the study and for 24 months after discontinuation of Vismodegib
14. Agreement not to donate blood or blood products during the study and for at least 24 months after discontinuation of Vismodegib.
15. Life expectancy > 12 weeks
16. Patients covered by a Health Insurance System

Exclusion Criteria:

1. Inability or unwillingness to swallow capsules
2. Patients with BCC situated out of the head or the neck area
3. Pregnancy or lactation
4. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy or photodynamic therapy
5. Chemotherapy within 4 weeks prior to enrollment
6. Participation in another clinical trial within 4 weeks prior to enrollment
7. Radiotherapy within 6 months prior to enrolment
8. Metastatic BCC
9. Uncontrolled medical illnesses such as infection requiring treatment with intravenous antibiotics.
10. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or that renders the patient at high risk from treatment complications.
11. Patients with a rare hereditary problem of galactose intolerance, primary hypolactasia or glucose-galactose malabsorption (according to the product SmPC).
12. Patients unable or unwilling to comply with the protocol requirements
13. Patients in emergency situations
14. Patients kept in detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
the change in surgery stages | Between baseline and maximum 10 months of treatment
  comparison of the surgery stages before and after the treatment with Vismodegib according to specific surgery stage table

SECONDARY OUTCOMES:
Number of patients with locally advanced BCC with down-staging of surgical procedures with Vismodegib | from 4 to 10 months of treatment
Gravity index related to the surgical or functional results (global score) | At maximum 10 months of treatment
Score of the clinical benefits at BOR | At maximum 10 months of treatment
Assessment of treatment toxicity according to NCI-CTC, v4.0 | 2 months after the surgery and maximum 12 months after the Vismodegib initiation
  National Cancer Institute - CommonToxicity Criteria (NCT-CTC) for the recognition and grading severity of adverse effects of chemotherapy
Quality of life assessment by Skindex-16 questionnaire | At screening, at 3 months, at 6 months of treatment
the tumor recurrence rate | at 3 years of follow-up
the cytological response by biopsy | from 4 to 10 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MORTIER, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (17):
- France (17):
  - CHU de Besançon, Besançon
  - Hôpital St André, Bordeaux
  - CH de Boulogne sur mer, Boulogne-sur-Mer
  - CHU - Hôpital d'Estaing, Clermont-Ferrand
  - CHU Bocage, Dijon
  - Clinique de Dermatologie, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Saint Eloi, Montpellier
  - Hôpital Bichat, Paris
  - Hôpital Saint-Louis, Paris
  - CHU Ambroise Paré, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Robert Debré, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No